CLINICAL TRIAL: NCT04443543
Title: Watch and Wait Strategy in Patients With Locally Advanced Rectal Cancer After Neoadjuvant Chemoradiotherapy: A Multi-centre, Adaptive-design, Phase II Prospective Cohort Study
Brief Title: An Adaptive-design Prospective Cohort Study of Watch and Wait Strategy in Patients With Locally Advanced Rectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhu Ji, principle investigator, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CARTOnG-2001
Record Dates: First submitted 2020-06-20; First posted 2020-06-23 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Rectal Cancer
Keywords: Chemoradiotherapy; organ preservation; watch and wait; irinotecan; Tislelizumab; capecitabine
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Irinotecan; Oxaliplatin; Fluorouracil; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Arm 1 includes patients with MSS/pMMR. In this arm, patients receive consolidation chemotherapy after neoadjuvant chemoradiation (nCRT). The chemotherapy regimens either XELIRI or FOLFIRINOX, and the cycles of chemotherapy depend on patient tumor responses. For patients who reach cCR will enter the "W&W" cohort and omit radical surgery, while those without cCR will receive radical surgery.
  Interventions: Drug: Capecitabine (Xeloda) Pharmacogenetic Test Reagents; Drug: irinotecan; Radiation: IMRT; Drug: Oxaliplatin; Drug: 5Fluorouracil
- Arm 2 (Experimental): Arm 2 includes patients with MSI-H/dMMR status. In this arm, patients receive consolidation immunotherapy of 3 cycles of tislelizumab after nCRT. For patients who reach cCR will enter the "W&W" cohort and omit radical surgery, while those without cCR will receive radical surgery.
  Interventions: Drug: Capecitabine (Xeloda) Pharmacogenetic Test Reagents; Drug: irinotecan; Radiation: IMRT; Drug: Tislelizumab

INTERVENTIONS:
Drug: Capecitabine (Xeloda) Pharmacogenetic Test Reagents — CRT: 625mg/m2 bid Monday-Friday per week XELIRI: 1000mg/m2 bid d1-14
Drug: irinotecan — CRT:80mg/m2 (UGT1A1*28 6/6) or 65mg/m2 (UGT1A1*28 6/7) XELIRI: 200mg/m2 bid d1 FOLFIRINOX: 150mg/m2 d1
Radiation: IMRT — Pelvic Radiation: 50Gy/25Fx
Drug: Oxaliplatin — FOLFIRINOX: 85mg/m2 d1
  Arms: Arm 1
Drug: 5Fluorouracil — FOLFIRINOX: 400mg/m2 iv d1bolus, 2400mg/m2 ivgtt 46h
  Arms: Arm 1
Drug: Tislelizumab — 200mg iv
  Arms: Arm 2

SUMMARY:
The study is designed to test the hypothesis that the clinical complete response (CCR) rate of patients with locally advanced rectal cancer (LARC) treated with neoadjuvant chemoradiotherapy will increase after an adaptive-design paradigm, as well as the rate of 2-year organ preservation, recurrence, quality of life, DFS and OS.

DETAILED DESCRIPTION:
1. Primary objective:

   Evaluate the CCR rate of low rectal cancer using adaptive and optimized chemotherapy and radiotherapy strategies (all population and dMMR/MSI-H subgroup)
2. Secondary objectives:

   2.1 Evaluate the 2-year anal preservation rate, recurrence rate, quality of life, DFS and OS 2.2 Explore the subgroup of patients suitable for observation.
3. Outline:

Patients after long-course chemoradiation are grouped based on their MSI-H/dMMR status. For patients with MSI-H/dMMR, consolidation immunotherapy of Tislelizumab (BGB-A317) will be assigned. For patients with MSS/pMMR, consolidation chemotherapy will be given according to their tumor response. After completion of consolidation therapy, those who reach clinical complete response will receive organ preservation (watch and wait) strategy in place of radical surgery. During treatment, once local regrowth occurs or poor tumor response, total mesorectal excision (TME) surgery will be performed.

ELIGIBILITY:
Inclusion Criteria:

* pathological confirmed adenocarcinoma
* clinical stage T2-4 and/or N+, inappropriate for local excision
* the distance from anal verge less than 5 cm, or considered inappropriate for anal preservation by surgeons.
* Strong desire to preserve the anus, able to receive close surveillance for at least 2 years after chemoradiotherapy.
* without distance metastases
* aged between 18 to 75 years old.
* performance status score: 0~1
* UGT1A1*28 6/6 or 6/7
* sign the inform consent

Exclusion Criteria:

* pregnancy or breast-feeding women
* serious medical illness
* difficult to achieve complete response assessed by current evidence: the maximal diameter of tumor >10cm; the maximal diameter of lateral lymph node >2cm; baseline CEA>=100; biopsy pathology confirmed signet ring cell carcinoma components; digital rectal examination found that the tumor is peri-narrowed.
* baseline blood and biochemical indicators do not meet the following criteria: neutrophils≥1.5×10^9/L, Hb≥90g/L, PLT≥100×10^9/L, ALT/AST ≤2.5 ULN, Cr≤ 1 ULN
* DPD deficiency
* UGT1A1*28 7/7

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2020-06-22 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
clinical complete response rate | two weeks after completion of CRT or consolidation chemotherapy.
  After nCRT, the lesions of rectal completely respond. Tumor residue cannot be found by digital rectal examination, endoscopic biopsy and radiology.

SECONDARY OUTCOMES:
2y-anal preservation rate | 2 years
  2-year anal preservation rate will be defined as the percentage of patients alive without receiving abdominoperineal resection at 2 years measured from the date of completion of CRT.
2y-local recurrence rate | 2 years
  2-year local recurrence rate will be defined as the percentage of patients alive developing local recurrence at 2 years measured from the date of completion of CRT.
Impact of participants' quality of life | 2 years
  quality of life is evaluated according to EORTC C-30 questionnare.
overall survival | 3 years
  3-year OS will be defined as the percentage of patients alive at 3 years measured from the date of completion of CRT.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Cencer, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No